CLINICAL TRIAL: NCT02985268
Title: Evaluation of Outcomes of Cardiac Resynchronization Therapy and MitraClip for the Treatment of Low Ejection Fraction and Functional Mitral Valve Regurgitation in Heart Failure
Brief Title: Evaluation of Outcomes of CRT and MitraClip for Treatment of Low Ejection Fraction and Functional Mitral Regurgitation in HF
Acronym: EVOLVE-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MHICC-2016-001
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Functional Mitral Regurgitation; Heart Failure
Keywords: MitraClip; Cardiovascular resynchronization therapy; Six minute walk test; Mitral regurgitation; CRT-D
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency | interventions — Cardiac Resynchronization Therapy; Defibrillators

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MitraClip/Optimal Medical Therapy (OMT) and CRT ON (Active Comparator): Patient to be implanted with both MitraClip and CRT-D. Will also receive optimal medical therapy. CRT-D will be programmed to ON
  Interventions: Device: MitraClip; Drug: Optimal Medical Therapy; Device: CRT-D
- MitraClip/OMT and CRT OFF (Active Comparator): Patient to be implanted with both MitraClip and CRT-D. Will also receive optimal medical therapy. CRT-D will be programmed to OFF until the 6-month follow-up visit in which the CRT will be turned ON
  Interventions: Device: MitraClip; Drug: Optimal Medical Therapy; Device: CRT-D
- OMT and CRT ON (Active Comparator): Patient to be implanted with only the CRT-D and will receive optimal medical therapy.
  CRT-D will be programmed to ON
  Interventions: Drug: Optimal Medical Therapy; Device: CRT-D
- OMT and CRT OFF (Active Comparator): Patient to be implanted with only the CRT-D and will receive optimal medical therapy.
  CRT-D will be programmed to OFF until the 6-month follow-up visit in which the CRT will be turned ON
  Interventions: Drug: Optimal Medical Therapy; Device: CRT-D

INTERVENTIONS:
Device: MitraClip — The MitraClip Clip Delivery System is indicated for the percutaneous reduction of significant symptomatic mitral regurgitation (MR ≥ 3+) due to primary abnormality of the mitral apparatus [degenerative MR] in patients who have been determined to be at prohibitive risk for mitral valve surgery by a heart team, which includes a cardiac surgeon experienced in mitral valve surgery and a cardiologist experienced in mitral valve disease, and in whom existing comorbidities would not preclude the expected benefit from reduction of the mitral regurgitation.
  Arms: MitraClip/OMT and CRT OFF; MitraClip/Optimal Medical Therapy (OMT) and CRT ON
Drug: Optimal Medical Therapy — Optimal medical therapy administered as per the Guideline Direct Medical Therapy (GDMT) as defined in the 2013 ACCF/AHA Heart Failure Guidelines with maximum tolerated doses of an ACE-inhibitor or Angiotensin Receptor Blocker (ARB) and beta-blocker
  Other Names: OMT
Device: CRT-D — Cardiac Resynchronization Therapy with defibrillation therapy devices will be implanted according to the Heart Rhythm Society Guidelines for implanted devices.
  Other Names: Cardiac Resynchronization Therapy and Defibrillator

SUMMARY:
At present, the optimal treatment strategy for heart failure patients and moderate-to-severe (3+) or severe (4+) mitral regurgitation with a class IIa recommendation for CRT is uncertain.Whether these patents should also be treated for functional mitral regurgitation or with CRT also remains unclear. We therefore propose a randomized 2x2 factorial design in this patient population to understand the the impact of both CRT and transcatheter mitral valve repair with the MitraClip on their functional status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic moderate-to-severe (3+) or severe (4+) functional mitral regurgitation due to cardiomyopathy of either ischemic or non-ischemic etiology as determined by transthoracic echocardiogram (TTE), and confirmed by the Echocardiography Core Lab (ECL);
2. Symptomatic heart failure as defined by New York Heart Association (NYHA) class II, III or ambulatory IV;
3. Treatment and compliance with optimal medical therapy for heart failure for at least 30 days; Optimal medical therapy is defined by: Maximum tolerated beta-blocker, angiotensin converting enzyme inhibitor (ACE) or angiotensin receptor blocker (ARB), and aldosterone antagonist (as per the ACCF/AHA Guidelines as judged by the HF specialist investigator on site and confirmed by the Clinical Eligibility Committee).
4. Left ventricular ejection fraction ≤ 35%, as assessed by any one of the following methods: echocardiography, contrast left ventriculography, gated blood pool scan or cardiac magnetic resonance imaging (MRI);
5. Class IIa indication for cardiac resynchronization therapy:

   1. Left bundle branch block (LBBB) and QRS duration of 120-149 ms;
   2. Right bundle branch block (RBBB) and QRS ≥ 150 ms.
6. Clinical agreement amongst local investigators that the patient will not be offered surgical intervention;
7. The primary regurgitant jet, in the opinion of the MitraClip implanting investigator, can successfully be treated by the MitraClip. Treatment of commissural mitral regurgitation may be treated at the discretion of the operator. All major jets contributing the secondary MR will be treated with the MitraClip;
8. Ability to perform a six-minute walk test (6MWT) without substantial physical limitations and without use of a walker or wheelchair and distance walked in 6 minutes of ≤ 450m;
9. Ability and willingness to give written informed consent and to comply with the requirements of the study.

Exclusion Criteria:

1. Life expectancy less than 12 months due to noncardiac conditions;
2. ACC/AHA Stage D Heart Failure;
3. Left ventricular ejection fraction ≤ 15%;
4. Hypotension (systolic pressure <90 mm Hg) or requirement for inotropic support or mechanical hemodynamic support;
5. United Network for Organ Sharing (UNOS) status 1 heart transplantation or prior orthotopic heart transplantation;
6. Untreated clinically significant coronary artery disease requiring revascularization;
7. CABG within prior 30 days;
8. Percutaneous coronary intervention within prior 30 days;
9. Severe Chronic Obstructive Pulmonary Disease (COPD) requiring continuous daytime home oxygen or chronic oral corticosteroid therapy;
10. Previous surgical mitral valve bioprosthesis, mitral annuloplasty, or transcatheter mitral valve procedure;
11. Positive pregnancy test, or woman of child bearing potential not using highly effective methods of contraception;
12. Mitral valve area <4.0 cm2 as assessed by planimetry of the mitral valve;
13. Subjects in whom trans-esophageal echocardiography is contraindicated or high risk;
14. Mitral leaflet anatomy which may preclude MitraClip implantation:

    1. Perforated mitral leaflets or clefts, lack of primary or secondary chordal support;
    2. Severe calcification in the grasping area;
    3. Rheumatic valve disease.
15. Previously implanted Cardiac Resynchronization Therapy and Defibrillator (CRT-D) system;
16. Stroke or transient ischemic event within 30 days before randomization;
17. Modified Rankin Scale >4 disability;
18. Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months;
19. Severe renal impairment defined as an Estimated Glomerular Filtration Rate (eGFR) <30 mL/min/1.73m2 as calculated by the Modification in Diet in Renal Disease (MDRD) formula;
20. Severe anemia requiring transfusional support or therapy with erythropoietin;
21. Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction;
22. Aortic valve disease requiring surgery or transcatheter intervention;
23. Significant tricuspid valve disease requiring surgical intervention or very severe tricuspid regurgitation;
24. Active infection requiring antibiotic therapy;
25. Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease;
26. Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
27. Any condition making it unlikely the patient will be able to complete all protocol procedures (including compliance with guideline directed medical therapy) and follow-up visits;
28. Presence of any of the following:

    1. Pulmonary artery systolic pressure (PASP) > 70 mm Hg confirmed by right heart catheterization;
    2. Infiltrative cardiomyopathies.
29. Any other condition(s) that would compromise the safety of the patient as judged by the site principal investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in distance walked on a six-minute walk test (6MWT) | Baseline to 6 months

SECONDARY OUTCOMES:
Change in cardiographic endpoints | Baseline to 6 months
  Mitral regurgitation severity
Change in cardiographic endpoints | Baseline to 6 months
  Indexed left ventricular end-systolic volume (LVESVi)
Change in cardiographic endpoints | Baseline to 6 months
  Left ventricular ejection fraction (LVEF)
Change in Quality of Life Assessment scores | Baseline to 6 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ)
Change in Quality of Life Assessment scores | Baseline to 6 months
  Euro Quality of Life Questionnaire (EQ5DL)
Number of Re-hospitalizations for decompensated heart failure | 6 and 12 months

OTHER OUTCOMES:
Wearable activity/heart rate sensor (Fitbit Charge 2) | 12 months
  Assessments obtained from the wearable activity/heart rate sensor:
  * Mean daily heart rate
  * Daily heart rate range calculated as the difference between min and max heart rate
  * number of daily steps
  * number of daily hours of sleep
Major Adverse Cardiac Event (MACE) | 12 months
  Time to major adverse cardiac events:
  * Cardiovascular death
  * All -cause mortality
  * non-fatal Myocardial Infarction
  * fatal and non-fatal stroke
  * rehospitalization for decompensated heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Anita Asgar, MD, Principal Investigator — Montreal Heart Institute

IPD SHARING:
Plan to Share IPD: No